CLINICAL TRIAL: NCT04241666
Title: Comparison of Sonographic Examination of Renal Function With Gold-standard Examination in Individuals With Long-term Spinal Cord Injury
Brief Title: Sonographic Examination of Renal Function in Individuals With Long-term Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Lotte und Adolf Hotz-Sprenger Stiftung (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-01
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries; Renal Insufficiency
MeSH Terms: conditions — Spinal Cord Injuries; Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- normal renal function: individuals with renal clearance >89 ml/min/1.73m²
  Interventions: Diagnostic Test: renal scintigraphy; Diagnostic Test: renal doppler sonography
- mild renal insufficiency: individuals with renal clearance 60-89 ml/min/1.73m²
  Interventions: Diagnostic Test: renal scintigraphy; Diagnostic Test: renal doppler sonography
- moderate renal insufficiency: individuals with renal clearance 30-59 ml/min/1.73m²
  Interventions: Diagnostic Test: renal scintigraphy; Diagnostic Test: renal doppler sonography

INTERVENTIONS:
Diagnostic Test: renal scintigraphy — Technetium-99m-dimercaptosuccinic acid scintigraphy of both kidneys
Diagnostic Test: renal doppler sonography — doppler ultrasound of both kidneys

SUMMARY:
Patients with long-term lower urinary tract dysfunction due to spinal cord injury presenting for a routine urodynamic control will be screened for inclusion and exclusion criteria. Suitable individuals providing written informed consent will undergo renal Doppler sonography and renal scintigraphy in addition to the routine examinations. Conclusions regarding renal function based on the clearance rate determined by scintigraphy (gold standard) will be compared with the conclusions based on Doppler sonography and Cystatin C clearance.

ELIGIBILITY:
Inclusion Criteria:

* long-term spinal cord injury (≥10 years)
* age ≥30 years
* written informed consent

Exclusion Criteria:

* dementia or severe intellectual impairment
* serious internal illness
* previous or current tumor disease
* known allergy to the radioactive marker (Technetium)
* pregnancy or breastfeeding
* withdrawal of informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with long-term lower urinary tract dysfunction due to spinal cord injury
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
renal clearance | at the time of inclusion into study
  renal clearance of Technetium-99m-dimercaptosuccinic acid determined by scintigraphy

SECONDARY OUTCOMES:
Cystatin C concentration | at the time of inclusion into study
  blood serum concentration of Cystatin C (mg/L)
Cystatin C clearance | at the time of inclusion into study
  renal clearance of Cystatin C (ml/min) according to the Grubb formula
renal peak systolic velocity | at the time of inclusion into study
  Doppler sonography evaluation of renal blood flow during systolic heart phase (m/s)
renal peak enddiastolic velocity | at the time of inclusion into study
  Doppler sonography evaluation of renal blood flow during enddiastolic heart phase (m/s)
renal resistive index | at the time of inclusion into study
  (systolic velocity - enddiastolic velocity) / systolic velocity

OTHER OUTCOMES:
size of kidneys | at the time of inclusion into study
  size of kidneys evaluated by sonography
renal tissue echogenicity | at the time of inclusion into study
  renal tissue echogenicity evaluated by sonography
bladder evacuation method | at the time of inclusion into study
  method of bladder evacuation
lesion level | 1 year after spinal cord injury
  highest intact spinal cord segment
lesion severity | 1 year after spinal cord injury
  severity of spinal cord injury according to American Spinal Injury Association Impairment Score (AIS) (A = motor and sensory complete, B = motor complete and sensory incomplete, C & D = motor and sensory incomplete, E = motor and sensory intact)
duration of spinal cord injury | at the time of inclusion into study
  time from spinal cord injury to inclusion into study (years)
age | at the time of inclusion into study
  time from birth to inclusion into study (years)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wöllner, Dr., Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No
data will be made available upon reasonable request

REFERENCES:
- [Derived] Jehli E, Krebs J, Schirp U, Walter MA, Wollner J, Pannek J. Decoding kidney function: evaluating arterial resistive index and cystatin C serum values in individuals with spinal cord injury. World J Urol. 2025 Dec 15;44(1):43. doi: 10.1007/s00345-025-06135-w. PMID 41396487